CLINICAL TRIAL: NCT02172677
Title: ETUDE D'IMAGERIE PAR RESONANCE MAGNETIQUE FONCTIONNELLE CHEZ LE SUJET SAIN DES RELATIONS ENTRE MEMOIRE COLLECTIVE ET INDIVIDUELLE
Brief Title: The Influence of Collective Schemas on Individual Memory (MULTIBRAIN_1)
Acronym: MULTIBRAIN_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: La Région Basse-Normandie (Other); Université de Caen Normandie (Other); University Hospital, Caen (Other); Ecole Pratique des Hautes Etudes (Other); Equipement d'Excellence Matrice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C13-46; 2014-A00126-41 (Registry Identifier: ID RCB)
Record Dates: First submitted 2014-06-16; First posted 2014-06-24 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2017-10

CONDITIONS: Episodic Memory
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy participants (Experimental): Structural and functional MRI and memory assessment
  Interventions: Behavioral: Episodic memory task; Device: fMRI

INTERVENTIONS:
Behavioral: Episodic memory task
Device: fMRI

SUMMARY:
Schemas describe mental structures storing recurrent and organized pattern of information. Schemas may have a strong influence on the process of storing and retrieving new information into memory. Previous approaches in the cognitive neuroscience of memory have entirely focused on the individual dimension of preexisting schemas. In the real world though, much of our experiences and knowledge are collective or shared. Such social-cultural frameworks stored in collective memory may also reshape and reconfigure the construction of individual memories. Attempting to ascertain the influence of collective schema on the neural substrates of individual memories using cutting-edge brain imaging methods represents the challenge that MULTIBRAIN seeks to tackle. To achieve this goal, we will record brain activity in a group of 24 participants while there are remembering pictures from a tour at the World War II Memorial of Caen. This study will seek to identify brain areas of the prefrontal cortex encoding the organization of knowledge in collective memory using multivariate analyses of brain patterns of activation, and then to understand how such regions might modulate the recruitment of the hippocampus during episodic memory retrieval using analyses of effective connectivity. The organization of knowledge in collective memory is measured in parallel through 1) the analysis of French social memory of World War II using a corpus of 100 000 television and radio shows from the National Institute of Audiovisual, and 2) an internet task measuring the organization of individual knowledge in a large group of individuals that will allow to separate shared from non-shared memories of the World War II. Once collected, these data will help us to understand how collective schemas may reconfigure the organization of individual memories.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between 20 and 38 years old
* Affiliated to the French national health care system
* French native speaker
* Participated in a tour trip at the Memorial of Caen within the last 3 months
* Right-handed
* At least 2 years of education after graduating from high school
* Body mass < 30kg/m2
* Signed written consent form

Exclusion Criteria:

* Pregnancy or intent to get pregnant
* Person deprived of their liberty
* Person hospitalized without consent
* Minor
* Protected adults or people unable to give informed consent
* Person subjected to an exclusion period related to another protocol
* History of neurological or psychiatric disorders or existence of traumatic brain injury with loss of consciousness for more than one hour
* History of cancer with the last 5 years, excluding squamous cell carcinomas
* Alcoholism, antecedents of chronic alcoholism or drugs abuse
* Severe psychiatric disorders (according to DSM V diagnostic criteria) or psychological troubles which could affect participant's judgment
* Use of medication that may interfere with cognitive or cerebral functioning
* Presence of visual or hearing troubles that may compromise participant's ability to participate in the study
* MRI Contraindications

Ages: 20 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Blood Oxigen Level Dependent (BOLD) response as measured with fMRI | 1 hour

SECONDARY OUTCOMES:
Episodic memory performances - % of accuracy | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Viader, PUPH, Principal Investigator — University Hospital, Caen
Locations (1):
- GIP Cyceron, Caen, France

REFERENCES:
- [Background] Gagnepain P, Vallee T, Heiden S, Decorde M, Gauvain JL, Laurent A, Klein-Peschanski C, Viader F, Peschanski D, Eustache F. Collective memory shapes the organization of individual memories in the medial prefrontal cortex. Nat Hum Behav. 2020 Feb;4(2):189-200. doi: 10.1038/s41562-019-0779-z. Epub 2019 Dec 16. PMID 31844272